CLINICAL TRIAL: NCT06451497
Title: Phase 1 Dose Escalation Trial of ZM008, an Anti-LLT1 Antibody, as Single Agent Followed by Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Trial of ZM008 as Single Agent and in Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zumutor Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZM008-001
Record Dates: First submitted 2024-05-14; First posted 2024-06-11 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer; Esophageal Cancer; Head and Neck Squamous Cell Carcinoma; Pancreas Adenocarcinoma; Biliary Tract Cancer; Prostate Cancer; Urothelial Carcinoma; Colorectal Cancer; Triple Negative Breast Cancer; High Grade Ovarian Serous Adenocarcinoma; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Biliary Tract Neoplasms; Prostatic Neoplasms; Carcinoma, Transitional Cell; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Lymphoma, Large B-Cell, Diffuse | interventions — Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Dose escalation of ZM008.
  Interventions: Biological: ZM008

INTERVENTIONS:
Biological: ZM008 — Intravenous delivery
  Other Names: Antibody

SUMMARY:
This is a phase 1 dose escalation trial of ZM008, an anti-LLT1 antibody as a single agent followed by combination with Pembrolizumab in patients with advanced solid tumors who have exhausted all standard therapy available or are intolerant of the same.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years at the time of signing the informed consent form.
2. Patients with histologically confirmed diagnosis of locally advanced, locoregionally recurrent, not amenable to curative therapy, or metastatic solid tumors that have no standard therapeutic option or are intolerant to the therapies. Tumor types to be included are Non Small Cell Lung Cancer, Triple Negative Breast Cancer, Head & Neck Squamous Cell Cancer, Prostate Cancer, Colorectal cancer, pancreatic ductal adenocarcinoma, biliary tract cancer, high grade serous ovarian cancer, diffuse large B-cell lymphoma or Urothelial Cancer.
3. Patients with tumors with actionable mutations should have progressed on all approved targeted therapies or have them contraindicated.
4. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 on computed tomography (CT), positron emission tomography (PET)/CT or magnetic resonance imaging (MRI) scan.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
6. The patient has adequate hematologic function as defined by:

   * Hemoglobin ≥9 g/dL (whole or partial blood transfusions not allowed in the weeks).
   * Absolute neutrophil count ≥1.0 × 109/L (growth factors like granulocyte colony- stimulating factors are not allowed in the two previous weeks).
   * Platelet count ≥75 × 109/L (platelet transfusions are not allowed in the 2 previous weeks).
7. The patient has adequate hepatic function as defined by:

   * Total bilirubin ≤1.5 times upper limit of normal (ULN).
   * AST and ALT ≤3.0 times ULN, (if liver metastases are present, then ≤5.0 times ULN is allowed).
8. The patient has adequate renal function as defined by:

   • Estimated creatinine clearance (CrCL) using the Cockcroft-Gault formula

   ≥30 mL/minute. Patients with calculated CrCL <30 mL/minute can be enrolled if measured CrCL is ≥30 mL/minute.
9. Women of childbearing potential (WOCBP) and men with sexual partners who are WOCBP must consent to adhere to contraceptive requirements from the day of the signature of the informed consent to at least 4 months after the last dose of trial treatment.
10. Suitable venous access for safe drug administration and the trial-required drug concentration and pharmacodynamic sampling.
11. Access to archival biopsy if available. If no archival tissue is available, the patient can still be enrolled in the escalation phase but not in the subsequent cohort expansion study. Part 2.

Exclusion Criteria:

1. Patients should have recovered from toxicity related to previous anticancer treatments (including surgery and radiation) to Grade 0/1 or baseline (except alopecia and peripheral neuropathy). Patients with endocrinopathies should have stable replacement treatment.
2. The patient has a history of uncontrolled brain metastasis. Patients with brain metastases are allowed if they are previously treated with surgery, whole-brain radiation, or stereotactic radiosurgery and have new brain imaging confirming that brain metastasis are stable (without evidence of progression by imaging using the identical imaging modality for each assessment, either MRI or CT) and considered controlled with <10 mg/day prednisone equivalent at the time of receiving the first dose of ZM008.
3. The patient has received extended field radiotherapy ≤4 weeks before the start of treatment (≤2 weeks for limited field radiation for palliation), and who has not recovered to Grade ≤1 or baseline from related adverse effects of such therapy (except for alopecia).
4. An active infection requiring parenteral or oral antibiotics at the time of the first dose. Oral antibiotics may be allowed if patient stable.
5. The patient has evidence of serious uncontrolled medical disorder that, in the opinion of the investigator or Medical Monitor, makes it unwise for the patient to participate in the trial or that might jeopardize compliance with the protocol.
6. The patient has a psychiatric illness/social circumstance that would limit compliance with trial requirements and substantially increase the risk of AEs or has compromised ability to provide written informed consent.
7. The patient has clinical evidence of an active second invasive malignancy with the exception of stable Prostate Cancer on watchful waiting, in situ cervical cancer, in situ breast carcinoma or localized non-melanoma skin cancers.
8. The patient has uncontrolled or significant cardiovascular disease defined as New York Heart Association classification III or IV.
9. The patient has baseline QTc (using the Fridericia correction calculation) >470 msec in patients without pacemaker.
10. The patient has history of autoimmune disease requiring systemic immunosuppressive therapy (daily prednisone equivalent doses >10 mg/day) excluding vitiligo, type I diabetes, Grave's disease, or Hashimoto thyroiditis.
11. Patients who discontinued prior treatment with any immune checkpoint due to immune-related AEs, irrespective of grade, recovery, or need for continued steroid therapy. Also, patients without formal contraindication due to previous irAE are not eligible if the AE has not resolved to Grade 1 or better and/or still requires steroids (>10 mg of prednisone equivalent per day) for ongoing management.
12. Patients has history of pneumonitis/interstitial lung disease due to any cause (infection, secondary to other treatments or idiopathic).
13. The patient has live vaccines reception within 30 days of enrollment.
14. Known active hepatitis B or C.
15. Patients positive for human immunodeficiency virus (HIV) can be enrolled only in the Part 2 of the trial, but HIV-positive patients must meet the following criteria:

    1. have CD4+ T cell (CD4+) counts ≥350 cells/μL.
    2. have not had an opportunistic infection within the past 12 months. Patients on prophylactic antimicrobials can be included in the trial.
    3. should be on established antiretroviral therapy for at least 4 weeks.
    4. have an HIV viral load of less than 400 copies/mL prior to enrollment.
    5. known history of any other relevant congenital or acquired immunodeficiency other than HIV infection.
16. Has known or suspected allergy to trial treatment, excipients, or related products.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Nature and frequency of dose limiting toxicities per Common Toxicity Criteria for Adverse Events version 5 | This starts at the beginning of screening procedures and upto 90 days after completion of the last cycle of investigational product administration with each cycle of 21 days duration.
  Adverse Events to be assessed.
Change in systolic and diastolic BP, | During screening (baseline), through the administration of investigational product (Day1 of each treatment cycle which is 21 days), end of treatment visit which is 30 days after completion of the last treatment cycle.
  Systolic & Diastolic measurements will be in mmHg
Change in Heart Rate | During screening (baseline), through the administration of investigational product, (Day1 of each treatment cycle of 21 days duration), end of treatment visit at 30 days after completion of last cycle of investigational product.]
  This will be measured in beats per minute.
Changes in Temperature measurements. | During screening (baseline), through the administration of investigational product, (Day1 of each treatment cycle of 21 days duration), end of treatment visit at 30 days after completion of last cycle of investigational product.]
  This will be measured in degrees Fahrenheit

SECONDARY OUTCOMES:
Overall Response Rate (ORR) per RECIST 1.1 | Assessed at study completion in upto 36 months.
  This calculation is defined as the percentage of patients with partial response (PR) or complete response (CR) per Response Evaluation Criteria in Solid Tumors (RECIST)1.1 version 5 based on local investigator assessment.
Immune Overall Response Rate (iORR) per iRECIST | Assessed at study completion in upto 36 months.
  This calculation is defined as the percentage of patients with partial response (PR) or complete response (CR) per Response Evaluation Criteria in Solid Tumors i(RECIST).
Progression Free Survival | From the start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  This is defined as the start of study treatment until disease progression per RECIST 1.1 or death from any cause for patients that have not started any other treatment for tumor reduction.
Immune Progression Free Survival | From start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  This is defined as the start of study treatment until disease progression per iRECIST or death from any cause for patients that have not started any other treatment for tumor reduction.
Disease Control Rate | From start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  This is defined as the percentage of patients with Complete Response, Partial Response and Stable Disease per RECIST criteria 1.1
Immune Disease Control Rate | From the start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  This is defined as the percentage of patients with Complete Response, Partial Response and Stable Disease per iRECIST criteria
Immunogenicity of ZM008 | Baseline, and before every cycle of investigational product administration (with each cycle being 21 days duration) and 30 days after last cycle completion.
  Blood will be drawn for antibodies against ZM008
Maximum Plasma Concentration of the biological product ZM008 | Baseline, on Cycle 1 Day1 (before and end of ZM008 infusion, 2 hour, 6 hour, 10 hour and 24 hour after infusion), day 2, day 8 & day15. Blood tests will be repeated for Cycle 2. Cycle 3 &4 onwards only Day 1 blood will be drawn. Cycle duration is 21 days
  Blood will be drawn for evaluating the maximum plasma concentration in micrograms/milliliter
Area Under the Plasma Concentration Versus Time Curve (AUC) of the biological product ZM008 | Baseline, on Cycle 1 Day1 (before and end of ZM008 infusion, 2 hour, 6 hour, 10 hour and 24 hour after infusion), day 2, day 8 & day15. Blood tests will be repeated for Cycle 2. Cycle 3 &4 onwards only Day 1 blood will be drawn. Cycle duration is 21 days
  Blood will be drawn at periodic intervals and the measure expressed as microgram/milliliter versus time in hours

CONTACTS AND LOCATIONS:
Overall Officials: Maloy Ghosh, PhD, Study Chair — Zumutor Biologics Inc.; Jyotsna Fuloria, Study Director — Fuloria Clinical Research Solutions LLC
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - NEXT Oncology, Austin, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No